CLINICAL TRIAL: NCT03772379
Title: Evaluation of Rapid Maxillary Expansion Facilitated by Micro-osteoperforation in Adolescent Patients With Skeletal Maxillary Constriction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mennatallah Ihab Elsayed, researcher assisstant at the national research center, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PhD Protocol
Record Dates: First submitted 2018-11-27; First posted 2018-12-11 (Actual); Last update posted 2018-12-11 (Actual); Status verified 2018-12

CONDITIONS: Posterior Crossbite

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tooth borne hyrax expander group (Experimental): patients of this group will receive a tooth borne hyrax expander anchored to the first premolars and first permanent molars .
  Interventions: Device: tooth borne hyrax expander
- tooth borne hyrax expander with microosteoperforation (Experimental): patients of this group will receive a tooth borne hyrax expander anchored to the first premolars and first permanent molars and microosteoperforation .
  Interventions: Procedure: microosteoperforation

INTERVENTIONS:
Device: tooth borne hyrax expander — ready made four stainless steel bands will be supported on the first premolars and first permanent molars and to which the palatal expander will be soldered to form the Hyrax,.The appliance will be activated one quarter turn per day untill reaching maximum amount of lateral expansion of the jack screw. the patients will be recalled twice per week to evaluate the progress of treatment.
  Arms: tooth borne hyrax expander group
Procedure: microosteoperforation — ready made four stainless steel bands supported on the first premolars and first permanent molars and to which the palatal expander will be soldered to form the Hyrax.No activation will be provided to the hyrax expander before the micro-osteoperforation is performed.
  Microosteoperforation will applied bilaterally on the buccal surface between the roots of teeth at the level of mucoginival junction, starting from the distal of canine till the distal of the first permanent molar using a small sized surgical bur mounted on a hand piece .
  Arms: tooth borne hyrax expander with microosteoperforation

SUMMARY:
The aim of this study is to evaluate and compare the effect of rapid maxillary expansion with and without microosteoperforation in patients with skeletal maxillary constriction.Theoretically, the force generated by the activation of the Hyrax expander leads initially to the compression of the periodontal ligament, bending of the alveolar bone, and tipping of the anchor teeth. This in turn contributes to the unfavorable changes in the supporting tissues; such as root resorption, buccal crown tipping, reduction of buccal bone thickness, marginal bone loss and alveolar bone fenestration and dehiscence. In this trial, it is assumed that by reducing the cortical bone resistance, using micro-osteoperforation (MOP), the alveolar bone bending and buccal tipping that usually occur during expansion will be reduced and thus facilitating the bone expansion.

DETAILED DESCRIPTION:
The study consists of 2 groups that are divided divided equally and randomly.The first group will receive a tooth borne Hyrax expander supported on first premolar and first permanent molar , whereas the second group will receive the same appliance associated with microosteoperforation(MOP). The MOP will be performed on the buccal segment bilaterally along the maxilla starting from the distal of the canine till the distal of the first permanent molar. The assessment will be done using CBCT scans immediately after expansion and 6 months postretention.

ELIGIBILITY:
Inclusion Criteria:

* Female adolescent patients with an age range 11- 14 years.
* Having apical constricted maxillary arch reflected by posterior cross-bite and verified through Howe's analysis on the dental study models.
* Normal vertical growth pattern.
* Fully erupted maxillary first premolars and first permanent molars.

Exclusion Criteria:

* Previous orthodontic treatment.
* Any congenital anomalies, systemic disease, or asymmetries that might have an influence on tooth movement.
* Active periodontal affection or severe gingival inflammation.

Ages: 11 Years to 14 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 34 (Estimated)
Dates: Start 2019-02 (Estimated); Primary Completion 2020-02 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Dental tipping. | an average1 year
  it will be measured in degree on Cone beam computed tomography image using a software
Alveolar bending | an average1 year
  it will be measured in degree on Cone beam computed tomography image using a software
Dental changes(transverse). | an average1 year
  it will be measured in mm on Cone beam computed tomography image using a software
Skeletal changes(transverse, anteroposterior and vertical) | an average1 year
  it will be measured in mm on Cone beam computed tomography image using a software

SECONDARY OUTCOMES:
Pattern of expansion | an average1 year
  it will be assessed on Cone beam computed tomography image and in mm clinically with boley gauge.